CLINICAL TRIAL: NCT03930589
Title: A Multi-center Randomized Trial of Remote Ischemic Conditioning to Reduce Infarct Size in Patients With an ST-Elevation Myocardial Infarction
Brief Title: Remote Ischemic Conditioning in STEMI to Decrease Infarct Size
Acronym: RemCon-STEMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Canadian VIGOUR Centre (Other)
Responsible Party: Principal Investigator, Robert Welsh, Professor, University of Alberta
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: V1 November 15, 2013
Record Dates: First submitted 2018-04-30; First posted 2019-04-29 (Actual); Last update posted 2019-04-29 (Actual); Status verified 2019-04

CONDITIONS: STEMI; CAD
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Remote ischemic condition versus standard of care
Who Masked: Outcomes Assessor
Masking Description: Patient outcomes and markers blinded to randomization arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care (Placebo Comparator): no intervention will occur in the standard of care arm
  Interventions: Other: Standard of care
- Remote Ischemic Conditioning (Active Comparator): Remote ischemic conditioning using BP cuff on left arm
  Interventions: Procedure: Remote Ischemic conditioning

INTERVENTIONS:
Procedure: Remote Ischemic conditioning — BP cuff inflation for 5 min and deflation for 5 mins with 4 cycles
  Arms: Remote Ischemic Conditioning
Other: Standard of care — Standard of care
  Arms: Standard of care

SUMMARY:
Following acute STEMI patients may have significant myocardial damage and subsequent heart failure. There is currently conflicting data regarding the benefit of remote ischemic conditioning to decrease the magnitude of infarction. Remote ischemic condition is a process where by repetitive intermittent limb ischemia is used to decrease the magnitude of myocardial damage caused by coronary artery occlusion and the subsequent reperfusion injury in STEMI patients. RemCon-STEMI is a multicenter randomized trial to test the impact of remote ischemic conditioning in acute STEMI.

ELIGIBILITY:
Inclusion Criteria:

Patients presenting with STEMI within 6 hours of symptom onset and:

1. Are expected to receive reperfusion therapy with either fibrinolysis or primary PCI.
2. Documented informed consent (verbal)

Exclusion Criteria:

1. Cardiogenic shock
2. History of anatomical deformity or vascular complication that limit ability to conduct remote ischemic preconditioning

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 251 (Actual)
Dates: Start 2013-11-08 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2018-11-26 (Actual)

PRIMARY OUTCOMES:
Composite of all cause death | 90 days
  all cause death, cardiogenic shock or chf through 90 days

SECONDARY OUTCOMES:
long term survival | up to 1 year
  survival
myocardial infarction size | within 72 hours of hospital admission
  mi size using peak elevation of cardiac biomarkers
ECG infarct size | with 10 days or hospital discharge whichever occurs first
  QRS score on baseline and discharge ECGS
Reperfusion | within 24 hours of admission to hospital
  ST segment resolution 30 minutes post PCI

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bainey KR, Zheng Y, Coulden R, Sonnex E, Thompson R, Mei J, Bastiany A, Welsh R. Remote ischaemic conditioning in ST elevation myocardial infarction: a registry-based randomised trial. Heart. 2022 May;108(9):703-709. doi: 10.1136/heartjnl-2021-319455. Epub 2021 Aug 20. PMID 34417205